CLINICAL TRIAL: NCT00856375
Title: A Multicenter, Open-Label, Randomized, Phase 2 Study to Evaluate the Efficacy and Safety of NKTR-102 Versus Irinotecan in Patients With Second-Line, Irinotecan-Naive, KRAS-Mutant, Metastatic Colorectal Cancer (mCRC)
Brief Title: NKTR-102 Versus Irinotecan in Patients With Second-Line, Irinotecan-Naïve, KRAS Mutant, Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-PIR-03
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Colorectal cancer, second line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — etirinotecan pegol; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NKTR-102 (Experimental): NKTR-102 IV every 3 weeks
  Interventions: Drug: NKTR-102
- irinotecan (Active Comparator): irinotecan IV every 3 weeks
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: NKTR-102 — IV every 3 weeks
  Other Names: etirinotecan pegol
  Arms: NKTR-102
Drug: irinotecan — IV every 3 weeks
  Arms: irinotecan

SUMMARY:
This study will evaluate whether NKTR-102, an investigational drug has an anti-tumor effect in patients with colorectal cancer. This study will also evaluate how the safety and anti-tumor activity of NKTR-102 compares with irinotecan, a cancer drug that is approved for use in the US for treatment of patients with certain types of colorectal cancer.

DETAILED DESCRIPTION:
NKTR-102 (Topoisomerase I Inhibitor Polymer Conjugate) is a polyethylene glycol (PEG) conjugate of irinotecan. Irinotecan is a topoisomerase I inhibitor approved worldwide. In the US, irinotecan is indicated as a component of first-line therapy in combination with 5 fluorouracil (5 FU) and leucovorin for patients with metastatic carcinoma of the colon or rectum. Irinotecan is also indicated for patients with metastatic carcinoma of the colon or rectum whose disease has recurred or progressed following initial fluorouracil-based therapy.

Second-line therapy for colorectal cancer typically involves cetuximab and irinotecan. However, growing evidence indicates that cetuximab (or other EGFR inhibitors) is not appropriate therapy for patients with mutant KRAS. For these patients, irinotecan may be appropriate as a single agent, and a new therapy that could improve upon efficacy and safety would provide an important option for the treatment of advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* metastatic colorectal cancer
* tumor with k-ras mutation

Exclusion Criteria:

* More than 1 prior regimen for treatment of metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-12; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (23):
- United States (9):
  - Investigator Site - Peoria, Peoria, Arizona
  - Investigator Site - Burbank, Burbank, California
  - Investigator Site - Los Angeles, Los Angeles, California
  - Investigator Site - Vallejo, Vallejo, California
  - Investigator Site - Centralia, Centralia, Illinois
  - Investigator Site - Louisville, Louisville, Kentucky
  - Investigator Site - Detroit, Detroit, Michigan
  - Investigator Site - Buffalo, Buffalo, New York
  - Investigator Site - Knoxville, Knoxville, Tennessee
- Investigator Site - Antwerp, Antwerp, Belgium
- Germany (2):
  - Investigator Site - Celle, Celle
  - Investigator Site - Karlsruhe, Karlsruhe
- India (7):
  - Investigator Site - Hyderabad, Hyderabad, Andhra Pradesh
  - Investigator Site - Ahmedabad, Ahmedabad, Gujarat
  - Investigator Site - Bangalore, Bangalore, Karnatak
  - Investigator Site - Kochi, Kochi, Kerata
  - Investigator Site - Mumbai, Mumbai, Maharashtra
  - Investigator Site - Kolkata, Kolkata, West Benagal
  - Investigator Site - Kolkata, Kolkata, West Bengal
- Spain (2):
  - Investigator Site - Elche, Elche
  - Investigator Site - Madrid, Madrid
- United Kingdom (2):
  - Investigator Site - Aberdeen, Aberdeen, Scotland
  - Investigator Site - Manchester, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- NKTR-102: NKTR-102 was administered as an intravenous (IV) infusion on Day 1 of each 21-day cycle at a dose level of 145 mg/m^2.
- Irinotecan: Irinotecan was administered as an IV infusion on Day 1 of a 21-day treatment cycle at a dose level of 350 mg/m^2. Patients aged 65 or older, or those with prior abdominal or pelvic irradiation, were given a lower dose of 300 mg/m^2.
Period: Overall Study
Arm/Group | NKTR-102 | Irinotecan
Started | 42 | 41
Completed | 0 | 0
Not Completed | 42 | 41
Not completed — Other | 0 | 1
Not completed — Death | 32 | 30
Not completed — Sponsor Terminated Study | 7 | 7
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Approximately 174 patients (87 patients per treatment arm) were originally planned to complete the trial. The study was terminated before completing accrual due to evolving standards of care with combination regimens that made recruitment to a Phase 2 study with single agent treatment difficult. Results of the 83 randomized patients (NKTR-102, n=42; irinotecan, n=41) were analyzed.
Groups:
- NKTR-102: NKTR-102
  NKTR-102: IV every 3 weeks
- Total: Total of all reporting groups
Arm/Group | NKTR-102 | Irinotecan | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.65) | 57.8 (11.4) | 58.2 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of PFS by Central Radiological Review: ITT Population
Description: PFS was defined as the time from the date of randomisation to the date of disease progression (assessed by central radiological review according to Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) or death due to any cause, whichever comes first. PFS was determined using the intention-to-treat (ITT) population which included all randomized patients who underwent baseline evaluation, with treatment assigned according to randomized arm. For patients whose disease did not progress or who did not die, the PFS time was censored at the time of the last tumor assessment that demonstrated lack of disease progression. For patients who received new anti-cancer therapy, the PFS time was censored at the time of last tumor assessment prior to the new anti-cancer therapy starts.
Time Frame: Every 6 weeks (± 5 days) from Cycle 1, Day 1 until documented disease progression, start of new therapy for cancer, death, or end of study, approximately 42 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NKTR-102 | Irinotecan
Number analyzed (Participants) | 42 | 41
months | 4.0 [2.7 to 5.9] | 2.8 [1.4 to 4.1]
Statistical Analysis 1: Comparison: NKTR-102 vs Irinotecan; Test type: Other — Hazard Ratio and 95% CI from univariate Cox regression model; p = 0.07, Log Rank; Hazard Ratio (HR) = 0.645, 95% CI 2-sided [0.4 to 1.041]

2. Secondary Outcome: Kaplan-Meier Estimate of OS: ITT Population
Description: Duration of OS was defined as the time from the date of randomization to the date of death due to any cause. Patients were followed until their date of death, loss to follow-up, withdrawal of consent for further follow-up for survival, or final database closure. Patients who were lost-to-follow-up or were not known to have died were censored at last date they were shown to be alive. Patients who did not have any follow-up since the date of randomization were censored at the date of randomization.
Time Frame: From randomization to death, loss to follow-up, withdrawal of consent for further follow-up for survival, or end of study, approximately 42 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NKTR-102 | Irinotecan
Number analyzed (Participants) | 42 | 41
months | 9.6 [7.3 to 13.2] | 8.4 [4.4 to 13.3]
Statistical Analysis 1: Comparison: NKTR-102 vs Irinotecan; Test type: Other — Hazard ratio and 95% CI from univariate Cox regression model; p = 0.706, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.557 to 1.486]

3. Secondary Outcome: ORR by Central Radiological Review: ITT Population
Description: ORR was defined as the proportion of patients with a complete response (CR) or a partial response (PR) per RECIST 1.1 based upon the best response as assessed by central radiological review; confirmation of response was not required. The analyses were performed for patients in the ITT population who had measurable disease as determined by the central imaging facility at baseline.
Time Frame: From randomization of the first subject until documented disease progression, start of new therapy for cancer, death, or end of study approximately 42 months
Measure: Median (95% Confidence Interval); unit: percentage of patients
Arm/Group | NKTR-102 | Irinotecan
Number analyzed (Participants) | 42 | 41
percentage of patients | 9.8 [2.7 to 23.1] | 5.0 [0.6 to 16.9]
Statistical Analysis 1: Comparison: NKTR-102 vs Irinotecan; Test type: Other — ORR 95% CI based on Exact (Clopper-Pearson) confidence limits. Odds ratio 95% CI based on asymptotic confidence limits; p = 0.676, Fisher Exact; Odds Ratio (OR) = 2.054, 95% CI 2-sided [0.355 to 11.9]

4. Secondary Outcome: DoR by Central Radiological Review: ITT Population
Description: Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that was the smallest on study); in addition to a relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. CR is defined as disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: From the time measurement criteria for CR/PR (whichever was first recorded) were first met until the first date that recurrent disease or PD or death was objectively documented, assessed until the end of study approximately 42 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NKTR-102 | Irinotecan
Number analyzed (Participants) | 42 | 41
months | 7.9 [1.5 to 11.6] | 1.4 [1.4 to 1.4]
Statistical Analysis 1: Comparison: NKTR-102 vs Irinotecan; Test type: Superiority; p = 0.018, Log Rank

5. Secondary Outcome: Percentage of Participants (≥2%) With Treatment-Emergent Adverse Events NCI-CTCAE Grade 3 or Higher
Description: An adverse event (AE) was any untoward medical occurrence in a patient administered a pharmaceutical product which did not necessarily have a causal relationship with the treatment. An AE could have been any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Pre-existing events, which increased in frequency or severity or changed in nature during or as a consequence of use of the study medication were also considered as AEs. All AEs were assessed for severity using the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3.0. If a particular AE was not listed in the NCI CTCAE Version 3.0, the following criteria were used: Grade 3 = severe; Grade 4 = life threatening or disabling; Grade 5 = death.
Time Frame: From the first dose of study medication through the End-of-Treatment visit (30 ± 3 days from last dose of study drug), assessed until the end of study approximately 42 months
Measure: Number; unit: % of participants
Arm/Group | NKTR-102 | Irinotecan
Number analyzed (Participants) | 42 | 41
% of participants
  Percentage of participants with ≥1 TEAE | 61.9 | 63.9
  Percentage of participants with Diarrhea | 21.4 | 19.5
  Percentage of participants with Neutropenia | 7.1 | 14.6
  Percentage of participants with Abdominal Pain | 14.3 | 4.9
  Percentage of participants with Dehydration | 9.5 | 9.8
  Percentage of participants with Vomiting | 11.9 | 7.3
  Percentage of participants with Nausea | 14.3 | 2.4
  Percentage of participants with Hypokalemia | 7.1 | 7.3
  Percentage of participants with Fatigue | 9.5 | 2.4
  Percentage of participants with Intestinal Obstruction | 2.4 | 9.8
  Percentage of participants with Leukopenia | 7.1 | 4.9
  Percentage of participants with Febrile Neutropenia | 2.4 | 7.3
  Percentage of participants with Alopecia | 2.4 | 4.9
  Percentage of participants with Disease Progression | 4.8 | 2.4
  Percentage of participants with Hyponatremia | 2.4 | 4.9
  Percentage of participants with Acute Prerenal Failure | 2.4 | 2.4
  Percentage of participants with Asthenia | 2.4 | 2.4
  Percentage of participants with Hyperbilirubinemia | 2.4 | 2.4
  Percentage of participants with Performance Status Decreased | 4.8 | 0
  Percentage of participants with Sepsis | 0 | 4.9

6. Secondary Outcome: PK Parameters of NKTR-102 or Irinotecan and Respective Metabolites
Description: Blood samples for PK analysis were collected from 4 patients only, 3 from the irinotecan treatment arm and 1 from the NKTR-102 treatment arm. NKTR-102, irinotecan, SN38, SN38-G, 7-ethyl-10-[4-N-(5-aminopentanoic acid)-1-piperidino]carbonyloxycamptothecin, and 7-ethyl-10-(4-amino-1-piperidino) carbonyloxycamptothecin concentration levels were determined. However, due to the limited number of patients with PK samples, no further PK analysis was conducted.
Time Frame: Days 1, 2, 3, 4, 8 and 15 of Cycles 1 and 3 and Day 1 of Cycles 2, 4 and all subsequent cycles, until End of Study, approximately 42 months.
Population: There are no data available for this outcome, due to the very small number of PK samples that were collected from these patients.
Arm/Group | NKTR-102 | Irinotecan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study medication through the End-of-Treatment visit (30 ± 3 days from last dose of study drug), assessed until the end of study approximately 42 months
Arm/Group | NKTR-102 | Irinotecan
All-Cause Mortality (participants affected / at risk) | 32/42 | 30/41
Serious Adverse Events (participants affected / at risk) | 19/42 | 24/41
Other Adverse Events (participants affected / at risk) | 42/42 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-102 (N=42) | Irinotecan (N=41)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 7 (8)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Diarrhoea Infectious (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (4) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-102 (N=42) | Irinotecan (N=41)
Haemoglobin decreased (Investigations) | 2 (7) | 6 (8)
Weight decreased (Investigations) | 13 (14) | 6 (6)
Neutrophil count decreased (Investigations) | 5 (8) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 6 (7) | 6 (7)
Leukopenia (Blood and lymphatic system disorders) | 5 (7) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 7 (14) | 5 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 4 (4)
Lethargy (Nervous system disorders) | 3 (10) | 5 (19)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 6 (10)
Vision blurred (Eye disorders) | 5 (5) | 1 (1)
Fatigue (General disorders) | 20 (25) | 18 (34)
Pyrexia (General disorders) | 4 (8) | 7 (7)
Asthenia (General disorders) | 6 (9) | 3 (4)
Oedema peripheral (General disorders) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 5 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 26 (62) | 28 (66)
Nausea (Gastrointestinal disorders) | 23 (41) | 24 (45)
Vomiting (Gastrointestinal disorders) | 17 (27) | 20 (33)
Abdominal pain (Gastrointestinal disorders) | 17 (25) | 13 (21)
Constipation (Gastrointestinal disorders) | 12 (18) | 10 (16)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 5 (5)
Proctalgia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (8) | 24 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 13 (15) | 10 (11)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (17) | 3 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.